CLINICAL TRIAL: NCT02009904
Title: Use of a Simple Breath Test to Examine Phenylalanine Metabolism in Children With Phenylketonuria (PKU)
Brief Title: Simple Breath Test to Examine Phenylalanine Metabolism
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Collaborators: Rare Disease Foundation, Vancouver, Canada (Other)
Responsible Party: Principal Investigator, Rajavel Elango, PhD, Principle Investigator, University of British Columbia
Other Study IDs: H12-01421
Record Dates: First submitted 2013-12-09; First posted 2013-12-12 (Estimated); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Phenylketonuria (PKU)
Keywords: PKU; Phenylketonuria; Phenylalanine; Children; Stable isotopes; Sapropterin dihydrochloride responsiveness
MeSH Terms: conditions — Phenylketonurias

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Breath samples from both groups (children with PKU and healthy controls)
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Phenylketonuria (PKU); Healthy Controls: Children with PKU (5-18y); Age and Gender matched healthy subjects for comparison

SUMMARY:
Phenylketonuria(PKU)is a rare condition caused by the body's inability to properly breakdown an amino acid called phenylalanine(PHE), due to a missing enzyme, phenylalanine hydroxylase(PAH). When the enzyme is missing and/or not functioning properly, it increases the level of PHE in the body. High levels of PHE can cause severe brain damage or nerve damage unless the children are on a strict low PHE diet. A low PHE diet restricts the intake of protein rich foods and can pose a significant burden to both the patient and the family.

Investigators at the University of British Columbia and British Columbia Children's Hospital will examine the phenylalanine metabolism in children with PKU using a simple breath test.

Patients (5-18y) receiving standard clinical care at the BC Children's Hospital's Biochemical Diseases Clinic will be enrolled.The study will be conducted twice on each patient. Baseline measurements will be performed at the beginning of each study for each patient.The Physician in charge will then prescribe the standard dose of sapropterin dihydrochloride (Kuvan®) (20mg/kg/d) or otherwise as deemed appropriate by the physician-in-charge. The test will be repeated a week (minimum) after the beginning of treatment with the prescribed dose.

The investigators propose that children who are responsive to sapropterin dihydrochloride (Kuvan®) will have increased 13CO2 in breath after treatment, and those who do not respond will have no change in the 13CO2 in the breath before and after treatment.

As a comparison to the experimental group, age and gender matched healthy controls will also be studied. The test in healthy controls will be performed once without any intervention, and is only used as a comparative value.

ELIGIBILITY:
Inclusion Criteria:

Study Subjects:

1. Children (4-18y)diagnosed with PKU
2. Parent(s) or guardian(s) willing and able to provide informed signed consent.
3. Parent(s) or guardian(s) willing and able to comply with all study procedures

Healthy controls:

1. Healthy Children (4-18y) with no health condition
2. Willing to go through an initial screening for age and gender match
3. Parents or guardians willing and able to provide informed signed consent.
4. Parents or guardians willing and able to comply with study procedures

Exclusion Criteria:

Study Subjects:

1. Children < 4y of age diagnosed with PKU, as it may be challenging to collect breath samples and perform indirect calorimeter in very young children
2. Children (4-18y)who are diagnosed with PKU, but are currently ill, with a fever, cold, vomiting or diarrhea

Healthy controls:

1. Healthy Children < 4y of age , as it may be challenging to collect breath samples and perform indirect calorimeter in very young children.
2. Healthy Children (4-18y), but are currently ill, with a fever, cold, vomiting or diarrhea.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children with PKU will be enrolled from the Biochemical Diseases clinic at the British Columbia Children's Hospital.
  Healthy controls will be enrolled from the community and will undergo screening for age and gender match.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2013-01; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
13C (carbon dioxide) production | 2 hours (1 study day)
  Breath samples are collected to measure 13C (carbon dioxide) production. Rate of carbon dioxide produced is measured at 60 minutes after the start of the study using an indirect calorimeter.

CONTACTS AND LOCATIONS:
Overall Officials: Rajavel Elango, Ph.D, Principal Investigator — University of British Columbia
Locations (1):
- Child & Family Research Institute, Vancouver, British Columbia, Canada